CLINICAL TRIAL: NCT02930317
Title: An Open-Label, Multicenter Evaluation of Safety, Pharmacokinetics, and Efficacy of rFVIII in the Prevention and Treatment of Bleeding Episodes in Chinese With Hemophilia A
Brief Title: Evaluate Efficacy and Safety of Recombinant Factor VIII （rFVIII）Treatment of Severe or Moderately Severe Hemophilia A
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTTQ-NXBYZ
Record Dates: First submitted 2016-09-09; First posted 2016-10-12 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmacokinetic parameters (Experimental): Pharmacokinetic parameters of rFVIII measured in subset of 10 participants, consisting of:18 Years to 65 Years. In Part 1 of the study, subjects received a single intravenous infusion of 50 IU/kg rFVIII preceded by a 72 hours washout period.
  Interventions: Drug: Recombinant Factor VIII (50 IU/kg)
- On-demand treatment (Experimental): On-demand treatment with rFVIII for 6 months age 12 Years to 65 Years. In Parts 2 of the study, subjects received repeat injections of rFVIII either as an on-demand or prophylaxis regimen at a dose and frequency determined by their study doctor.
  Interventions: Drug: Recombinant Factor VIII (On-demand treatment)

INTERVENTIONS:
Drug: Recombinant Factor VIII (50 IU/kg)
  Arms: Pharmacokinetic parameters
Drug: Recombinant Factor VIII (On-demand treatment)
  Arms: On-demand treatment

SUMMARY:
Efficacy, Safety and Pharmacokinetics Study of a rFVIII in Chinese subjects with Hemophilia A.To assess efficacy and safety of rFVIII administered as treatment and as on-demand therapy in adult and adolescent (12-65 years) patients with severe or moderately severe Hemophilia A. To determine the pharmacokinetic (PK) parameters of rFVIII.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hemophilia A
* Age of 12 Years to 65 Years，Diagnosis of severe （defined as <1% FVIII:C documented in medical records） or moderately severe（defined as 1%-5% FVIII:C documented in medical records） hemophilia A .Subjects who（Age of 18 Years to 65 Years） have received or are currently receiving FVIII products (plasma-derived and/or recombinant FVIII) and have had >150 exposure days (EDs) with a FVIII product；The Callan (Age of 12 Years to 17) have received FVIII products and have had>50 EDs a FVIII product.
* Subjects without a past history of, or current no factor VIII inhibitor. For laboratory-based assessments, any Bethesda inhibitor titer Lower than the laboratory's normal range or <0.6 BU/mL (BU:Bethesda Units ).
* Liver and kidney function in accordance with the standard
* Subjects of childbearing potential should agree to use and utilize an adequate method of contraception throughout treatment and for at least 28 days after study is stopped
* Evidence of a personally or legally acceptable representative (legally acceptable representative is only applicable to Callan subjects) signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study
* The part one of subjects subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures; Subjects must be in a non bleeding state before the administration of rFVIII on Day 1; Subjects should not have received an infusion of any FVIII products for at least 3 days (at least 72 hours) before the administration of rFVIII on Day 1

Exclusion Criteria:

* Current FVIII inhibitor or history of FVIII inhibitor (>0.6 BU/mL )
* Diagnosed with any bleeding disorder in addition to hemophilia
* Documented Human Immunodeficiency Virus (HIV)
* Subjects anticipating elective surgery or other invasive procedure within 1 month following study entry
* Treatment with an immunomodulatory within 30 days or 5 half lives preceding Day 1, whichever is longer
* Subjects with known hypersensitivity to the active substance or to any of the excipients of rFVIII. Subjects with a known hypersensitivity to Chinese Human embryonic kidney cell proteins
* Subjects with severe anemia requiring blood transfusion
* Subjects with significant hepatic or renal impairment (alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >5 x ULN, or total bilirubin >2 x ULN or serum creatinine >2 x ULN), prothrombin time >1.5 x ULN, platelet count <80,000 μL. History of sensitivity to heparin or heparin induced thrombocytopenia or others thrombocytopenia
* Patients with heart surgery history requires anticoagulation therapy; Subjects with severe heart disease, including myocardial infarction or heart failure Grade 3 or higher(NYHA Classification)
* Blood pressure unable to be controlled ideally(systolic pressure>150 mmHg，diastolic pressure>90 mmHg)
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Recovery rate = (change actual value of rFVIII activity before and after infusion )/(change expected value of rFVIII activity before and after infusion)*100% | At 15 and 60 minutes after the first infusion
Investigator Hemostatic Efficacy Assessment 6 Hours Post Infusion | 6 hours post infusion
  The Investigator Hemostatic Efficacy Assessment was based on a 4-point rating scale (Excellent = 1: definite pain relief or improvement in signs of bleeding, with no additional infusion, Good = 2: definite pain relief or improvement in signs of bleeding, Moderate = 3: probable or slight improvement, No Response = 4: no improvement at all between infusions).

SECONDARY OUTCOMES:
The proportion of subjects who achieved the expected effect after the first infusion of the rFVIII | At 15 minutes after the first infusion
change actual value of rFVIII activity before and after infusion levels | At 15 and 60 minutes after the first infusion
FVIII Maximum Plasma Concentration | Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 6, 9, 24,36,and 48 hours post-dose
Time to Reach Maximum Observed Plasma Concentration | Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 6, 9, 24,36,and 48 hours post-dose
Area Under the Plasma Concentration Versus Time Curve From 0 to 48 Hours | Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 6, 9, 24,36,and 48 hours post-dose
Terminal Elimination Half-Life (t1/2) | Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 6, 9, 24,36,and 48 hours post-dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 6, 9, 24,36,and 48 hours post-dose

OTHER OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs) | Up to 28 days after last dose
  An AE was any untoward medical occurrence in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose after last dose that were absent before treatment or that worsened relative to pre-treatment state. AEs included both SAEs and non-SAEs.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Anhui provincial hospital, Hefei, Anhui
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Second hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Blood Diseases Hospital, Chinese Academy of Medical Science (Institute of Hematology), Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Undecided